CLINICAL TRIAL: NCT04390035
Title: Blood Flow Restriction Training in the Adolescent Patient: Effects on Muscle Strength and Overall Function Following Anterior Cruciate Ligament Reconstruction Surgery
Brief Title: BFRT in Adolescents After ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Jeanne Perkis, Clinical Site Supervisor, Physical Therapist, Children's Healthcare of Atlanta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000434
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Adolescents; Blood Flow Restriction Training; Patient-reported Outcomes
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either a control group or the test group at time of enrollment at a 1:1 ratio. Participants will undergo standard post-surgery rehabilitation (control group) or standard post-surgery rehabilitation with supplemental blood flow restriction (test group).
Masking Description: Given that the intervention involves a device that will be physically applied to the participant's post-operative leg, masking is not feasible for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Participants in the control arm will follow the standard-of-care treatment exercises for the 6 months following ACL reconstruction surgery.
- Test (BFRT) (Experimental): Participants in the test arm will follow the identical physical therapy exercises as the control arm but will perform the exercises with BFRT during the first 16 weeks post-surgery. After reaching the 16-week mark, participants will complete the identical standard-of-care rehabilitation between weeks 16-24.
  Interventions: Device: Blood Flow Restriction using Delfi Personalized Tourniquet System

INTERVENTIONS:
Device: Blood Flow Restriction using Delfi Personalized Tourniquet System — Participants assigned to the test group will undergo blood flow restriction training 2 days per week beginning at week 1-2 post-surgery and continuing through week 16 post-surgery using the FDA-approved Delfi Personalized Tourniquet System (PTS) with personalized pressure of 80% of the limb occlusion pressure (LOP). The LOP is the amount of pressure required to fully occlude arterial and venous blood flow to the limb. Otherwise, both the test group and control group will follow a standard 6-month post-surgery rehabilitation protocol which is standard of care for ACLR recovery.
  Arms: Test (BFRT)

SUMMARY:
This is an interventional study that will examine effects of blood flow restriction training (BFRT) in adolescents aged 12-18 after anterior cruciate ligament reconstruction surgery (ACLR). The study aims to identify the effect of BFRT on quadriceps muscle strength and the patient's quality of life, and the overall tolerability of BFRT will be examined. Eight physical therapists at four sports medicine physical therapy (PT) sites will oversee all post-operative PT sessions. Subjects allocated to the BFR group will undergo BFRT, while control group will undergo standard-of-care ACLR rehabilitation, 2 days per week for 16 weeks. Measurements of strength, quality of life, and overall function will be completed at regular intervals.

DETAILED DESCRIPTION:
Background:

Approximately 100,000 anterior cruciate ligament reconstructions (ACLR) are performed yearly, and rates of these surgeries in patients younger than 15 years increased by 924% between 1990 and 2007.1 Persistent strength deficits in quadriceps musculature following ACLR are common, even several months after surgery and despite targeted physical therapy to address atrophy.2 Quadriceps atrophy and weakness are associated with worse patient-reported outcomes (PROs),3 as well as altered movement strategies and increased risk of reinjury.4,6 Approximately 20% of teenagers returning to sports will sustain a second ACL injury in the first two years following their ACLR.5 Regaining neuromuscular activation and strength of the quadriceps muscle safely and efficiently is vital to full recovery, and current post-operative physical therapy regimens have not sufficiently addressed this impairment.

Strength training models recommend utilizing high resistance workloads to produce substantial strength gains,7 yet those recovering from orthopedic surgery are unable to tolerate heavy loads.8 Supplementing low-load resistance training with blood flow restriction (BFR-LLT) produces significant muscle hypertrophy and strength gains previously only thought to be achievable with high-load resistance training.9 BFR-LLT uses a tourniquet around the leg (see Appendix 4) to partially occlude venous return and decrease blood supply to the muscle being exercised. The generation of a low-oxygen environment and increases in plasma growth hormone levels has been shown to promote recruitment of motor units, improve neuromuscular activation, and result in muscular hypertrophy and growth.10-13 In adults and the elderly, improvements in quadriceps strength have been reported in up to 19%14 and increased quadriceps cross-sectional area in up to 6-7% compared to controls.15-16 To date there have only been four high-level studies investigating effects of BFR training in patients following ACLR17-20 and limited conclusions can be drawn from these studies due to lack of consistent methodology (variable cuff pressures and treatment frequency). More high-quality research is needed to determine treatment parameters that produce the most optimal results from this intervention in ACLR patients.

Additionally, there are no published randomized controlled trials investigating the effects of BFR training on exclusively adolescent patients. All high-quality BFR training research in patients following knee surgery have been conducted in late adolescent, young adult and adult populations.17-21 Therefore, the purpose of this study is to assess the effect of BFR-LLT on quadriceps strength and outcomes in adolescents following ACLR.

This study's adolescent-specific focus provides a significant contribution to ACLR research, as younger patients demonstrate higher risk of reinjury.22-24 The results from this preliminary study will ultimately provide data to guide clinicians in optimizing quadriceps strength and utilizing BFR-LLT in younger post-operative ACLR patients.

Protocol:

This randomized clinical trial is an interdisciplinary project between the CHOA Sports Medicine Physical Therapy department and Children's Physician Group (CPG) Orthopedics. As part of standard-of-care, all patients who plan to undergo ACLR by CPG Orthopedics surgeons are referred for at least one PT visit pre-surgery, at which time baseline strength measurements are obtained by the treating physical therapist. Pre-surgery collection of patient-reported outcomes (PROs) is also standard of care for all patients undergoing ACLR.

Skeletally mature male and female adolescents with closed growth plates documented by radiograph who undergo ACLR with quadriceps tendon autograft will be screened by a physical therapist (the PI or co-investigators) using medical notes.

If a patient meets criteria and consents, he/she will be enrolled into the study during the first routine-of-care post-surgery PT visit and randomized to undergo standard post-surgery rehabilitation (control group) or standard post-surgery rehabilitation with supplemental BFR-LLT (test group) as demonstrated in Figure 1 and Appendix 1. Participants will be randomized using a computer program that will generate random numbers to assign participants to the test group or the control group. Participants will be asked to complete four PROs throughout the study (Lysholm, Pedi-IKDC, ACL-RSI, and AMCaMP - see Appendix 5.1-5.4). All relevant demographic, physiological, and radiographic data will be collected at the time of enrollment via RedCap, through a secure link. Data will be stored in a password-protected file on a secure Children's server and only the PI, Co-investigators, and research coordinator will have access.

Eight physical therapists (all CITI-trained) at four sports medicine PT sites will oversee all post-surgery PT sessions. Participants in the control group will follow a standard post-surgery rehabilitation protocol starting 2-5 days post-surgery and attend two PT visits per week until 16 weeks post-surgery. The test group will follow an identical schedule of PT visits but will have two to three exercises in each session supplemented with BFR treatment using the Delfi Personalized Tourniquet System (PTS). Requirements of BFR treatment are described below. For both groups, each session will last approximately 60 minutes. Each of the exercises performed with BFR will last 5-18 minutes, with total time under occlusion not exceeding 30 minutes per visit.

Participants undergoing BFR treatment will wear limb protection sleeves designed to help protect the skin beneath the cuff while the cuff is pressurized. Skin integrity will be monitored pre- and post-treatment at each session. If a study participant reports intolerable pain levels during BFR, the physical therapist will fully deflate the cuff and BFR treatment will cease for that PT session. Any adverse events will be reported to the PI and Co-I's within 24 hours. All required medical assessments will be promptly performed.

If a participant is assigned to the test group, BFR intervention will end after 16 weeks post-surgery. Both the test group (BFR-LLT) and the control group will follow standard of care treatment after week 16 post-surgery, including the standard post-intervention functional testing at 24 weeks post-surgery.

Participants will be asked to complete PROs periodically throughout the study as listed below under data collection. All physical examination measures and testing listed are standard of care for ACLR rehabilitation patients. Details on the regimen followed by both cohorts during the full 6-month rehabilitation are outlined in Appendix 1.

BFR-LLT Treatment Requirements:

The BFR-LLT intervention requires participants to follow the two requirements listed below, as the treatment parameter of 80% LOP has been widely recommended as the ideal amount of blood flow occlusion throughout the literature. Participants who do not meet these criteria will be excluded from the study but will continue to receive standard of care for post-surgery ACLR rehabilitation.

1. Tolerate a personalized pressure of 80% of the limb occlusion pressure (LOP) for 100% of all physical therapy visits in which BFR-LLT is utilized.
2. Tolerate BFR-LLT for a minimum of 20 visits over 16 weeks.

Data Collection:

1. Demographic data (pre-surgery, which is standard of care) will include age, gender, race/ethnicity, height/weight, physeal status, and assessment of baseline activity level with the Tegner Activity Scale (see Appendix 6)
2. Patient-reported outcomes (PROs) (see Appendix 5) will include the Pediatric Internal Knee Documentation Committee (Pedi-IKDC, Appendix 5.1), Lysholm Score (Appendix 5.2), ACL-Return to Sport after Injury (ACL-RSI) confidence assessment (Appendix 5.3) and Adolescent Measure of Confidence and Musculoskeletal Performance (AMCaMP,Appendix 5.4). These PROs are collected pre-surgery as standard of care, but further collection and reassessment of PROs as described in Figure 2 will be unique to study participants. Surveys will be collected and recorded on iPads with direct entry into REDCap and in each participant's confidential EHR on the treatment note from the day the data was collected. All responses will be stored on a secure RedCap server through a secure link and data will be stored in a password-protected file on a secure Children's server. Only the PI and Co-I's will have access to the data.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent male and female patients, age 12-18
2. Skeletally mature at time of diagnosis, with closed growth plates, as determined via standard clinic x-ray imaging (this specification automatically excludes pre-pubescent children.
3. Underwent transphyseal ACLR with quadriceps tendon autograft with one of three sports orthopedic surgeons at CHOA
4. Completed pre-surgery strength assessment of bilateral quadriceps, hamstrings, hip abductor and hip adductor musculature.
5. English-speaking adolescents and parents of all races and ethnicities (after preliminary data is achieved, PI will coordinate a larger multi-center study that will include all non-English speaking participants.

Exclusion Criteria:

1. Skeletally immature patients with open growth plates, as determined via standard clinic x-ray imaging
2. Concomitant procedures performed during ACLR which require weight-bearing restrictions (i.e. meniscus repair, microfracture, multi-ligament knee reconstruction)
3. History of previous knee surgery
4. History of cardiovascular disease (e.g. coronary artery disease, unstable hypertension, vascular endothelial dysfunction, peripheral artery disease, varicose veins)
5. ICD-10 diagnosis of bleeding disorder (e.g. hemophilia or blood clotting disorder) or use of anticoagulants or other medications that may affect blood clotting
6. Inability to adhere to treatment protocol (as described in study procedures, BFR-LLT treatment requirements)
7. Any adverse events intra-operatively or post-operatively that lead to delay in care, including infection
8. Failure to adhere to attendance requirements as detailed below:

   * Attend first PT visit (PTV) within 5 days post-surgery
   * Attend a minimum of 20 total PTVs during weeks 1-16 post-surgery

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Strength | 0-24 weeks post-surgery
  Quadriceps strength will be evaluated throughout the study using handheld dynamometry and percentage improvement will be compared between the control group and intervention group.
Hop Test Results | 24 weeks
  The hop test battery includes four hop tests (single leg hop for distance, triple hop for distance, 6-meter timed hop, triple crossover hop). Symmetry of performance between operative and non-operative lower extremity will be compared between control group and intervention group. The test will be performed at 24 weeks post-surgery.
Y-Balance Test Results | 24 weeks
  Symmetry of performance between operative and non-operative lower extremity will be compared between control group and intervention group. This test will be performed at 24 weeks post-surgery.

SECONDARY OUTCOMES:
Quality of life via Lysholm Knee Scale Score | At time of enrollment and 6, 12, and 24 weeks post-surgery
  The Lysholm Knee Scoring Scale is a patient-reported outcome which will be used to assess participant quality of life throughout the recovery following surgery. This tool asks eight questions and the score total ranges from 0-100 with 100 being the better outcome.
Discomfort during BFRT via Visual Analogue Scale | 0-16 weeks post-surgery
  The Visual Analogue scale is a patient-reported outcome, the score ranges from 0 - 10, with 0 being no pain. Pain level pre-treatment and during training will be assessed at each session
Perceived Exertion during BFRT via the Children's OMNI Resistance Training Scale. | 0-16 weeks post-surgery
  The children's OMNI resistance training scale is a patient-reported outcome, the score ranges from 0 - 10, with 0 being no exertion. Perceived exertion will be assessed at each treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Graf, PT, DPT, ATC, Principal Investigator — Clinical Site Supervisor, Physical Therapist
Locations (1):
- Children's Healthcare of Atlanta Physical Therapy, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.